CLINICAL TRIAL: NCT02634190
Title: Clinical Evaluation of the APTIMA® HPV Assay and Comparison With the HR HPV HC2® Test in Women 30 Years of Age or Older Using LBC ThinPrep® Pap Test Specimens
Brief Title: Clinical Evaluation of the APTIMA® HPV Assay and Comparison With the HR HC2® Test Using LBC ThinPrep® Specimens
Status: Completed | Type: Observational
Sponsor: Hologic Deutschland GmbH (Industry)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Aptima Study
Record Dates: First submitted 2015-12-03; First posted 2015-12-17 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Human Papilloma Virus Infection
Keywords: Cervical cancer screening; High risk Human Papillomavirus; Aptima HPV Assay
MeSH Terms: conditions — Papillomavirus Infections | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — liquid based cytology LBC Specimens (ThinPrep® Pap Test)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Triple negative women: Women 30 years of age or older coming for routine cervical screening who tested triple negative at baseline with the interventions: Thinprep® LBC, HR HC2® HPV DNA and APTIMA® HPV Assay
  Interventions: Other: Thinprep® LBC; Other: APTIMA® HPV Assay; Other: HR HC2® HPV DNA; Other: Colposcopy
- Women tested positive: Women who tested positive in any of the tests Thinprep® LBC, HR HC2® HPV DNA or APTIMA® HPV Assay will undergo colposcopy and be followed up over a ten year period and subjects who tested positive during the follow up assessment will be followed up over a 5 year period on a yearly basis
  Interventions: Other: Thinprep® LBC; Other: APTIMA® HPV Assay; Other: HR HC2® HPV DNA; Other: Colposcopy

INTERVENTIONS:
Other: Thinprep® LBC — liquid based cytology
Other: APTIMA® HPV Assay — in vitro diagnostic test
Other: HR HC2® HPV DNA — in vitro diagnostic test
Other: Colposcopy — Colposcopy

SUMMARY:
To assess and compare the performance of the HR HPV HC2® test (Qiagen/Digene) and the APTIMA® HPV Assay (Hologic) using LBC Specimens (ThinPrep® Pap Test) for the detection of HPV infection and high-grade CIN lesions in a screening population of women 30 years of age or older in Germany.

DETAILED DESCRIPTION:
The study is conducted in the areas of Tuebingen, Freiburg and Saarbruecken in Germany. In total, 10.000 ThinPrep® LBC cervical samples were collected from June 2009 to May 2012. Liquid based cytology (LBC) was performed by a central laboratory in Saarbruecken. Human papilloma virus (HPV) testing with the HR HPV HC2® test and APTIMA® HPV Assay were performed at the Section of Experimental Virology, Institute of Medical Virology, University Clinic of Tuebingen, Germany (UKT).

Within a follow-up phase women who tested positive in any test at baseline will be monitored over a period of 10 years.

Study close out visit: In addition, approximately 5 years after baseline ThinPrep® LBC cervical samples will be collected from a random sample of 4000 study participants who tested triple negative at baseline for determination of the longitudinal negative predictive value (NPV) and HPV related disease after a 5 year period. Women who tested positive in any test will undergo colposcopy.

ELIGIBILITY:
Inclusion criteria:

* Women aged 30 - 60 years
* Women attending gynaecological practices for routine screening
* Women who gave informed consent to participation in the study

Exclusion criteria:

* Women with hysterectomy or known destructive therapy to the cervix
* Women who are pregnant
* Women with an abnormal cytology result during the previous 6 months
* Women with known HIV infection or history of transplants
* Women vaccinated against HPV
* Women participating in another research protocol

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 30 years of age or older coming for routine cervical screening are enrolled in gynaecological practices.
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2009-06; Primary Completion 2021-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Overall high risk (HR) HPV prevalence with HR HC2® HPV and APTIMA® test | Baseline

SECONDARY OUTCOMES:
Sensitivity of LBC, HC2® and APTIMA® tests | Baseline, 5 years
Specificity of LBC, HC2® and APTIMA® tests | Baseline, 5 years
Positive Predictive Value (PPV) of LBC, HC2® and APTIMA® tests | Baseline
Negative Predictive Value (NPV) of LBC, HC2® and APTIMA® tests | Baseline
Prevalence of HR HPV infection by age with HC2® and APTIMA | Baseline, 5 years
Cross sectional association between HR HPV infection (HC2® and APTIMA) and LBC diagnosis | Baseline, 5 years
  Linear regression models will be used for determination of cross sectional associations between HR HPV Infection and LBC diagnosis.
Relative risk of cervical disease for positive tested women | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years
  Analysis of study results at baseline and follow-up visits. Calculation of relative risks of cervical disease for women who are positive for LBC, HC2® and/or APTIMA® test compared to those being negative for any of the three tests at the baseline visit.
Cumulative risk of cervical diseases for positive tested women at 5 years | Baseline, 1 year, 2 years, 3 years, 4 years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years

OTHER OUTCOMES:
Determination of longitudinal negative predictive value of HPV infection (HR HPV HC2® test or APTIMA® HPV or LBC) after a 5 year period | 5 years
  In triple negative study participants (HR HPV HC2® test and APTIMA® HPV and LBC) at baseline the longitudinal negative predictive value of HPV infections will be determined after a 5 year period.
Cumulative risk of Human Papilloma Virus (HPV) infection (HR HPV HC2® test or APTIMA® HPV or LBC) after a 5 year period | 5 years
  In triple negative study participants at baseline the cumulative risk of HPV infection will be determined after a 5 year period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Iftner, Prof., Principal Investigator — University Hospital Tuebingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iftner T, Becker S, Neis KJ, Castanon A, Iftner A, Holz B, Staebler A, Henes M, Rall K, Haedicke J, von Weyhern CH, Clad A, Brucker S, Sasieni P. Head-to-Head Comparison of the RNA-Based Aptima Human Papillomavirus (HPV) Assay and the DNA-Based Hybrid Capture 2 HPV Test in a Routine Screening Population of Women Aged 30 to 60 Years in Germany. J Clin Microbiol. 2015 Aug;53(8):2509-16. doi: 10.1128/JCM.01013-15. Epub 2015 May 27. PMID 26019212
- [Result] Iftner T, Neis KJ, Castanon A, Landy R, Holz B, Woll-Herrmann A, Iftner A, Staebler A, Wallwiener D, Hann von Weyhern C, Neis F, Haedicke-Jarboui J, Martus P, Brucker S, Henes M, Sasieni P. Longitudinal Clinical Performance of the RNA-Based Aptima Human Papillomavirus (AHPV) Assay in Comparison to the DNA-Based Hybrid Capture 2 HPV Test in Two Consecutive Screening Rounds with a 6-Year Interval in Germany. J Clin Microbiol. 2019 Jan 2;57(1):e01177-18. doi: 10.1128/JCM.01177-18. Print 2019 Jan. PMID 30355760